CLINICAL TRIAL: NCT01127945
Title: A Prospective, Single-center, Randomized, Controlled, Open-label, Pilot Study to Evaluate the Effectiveness of High Dose Statin Loading in Acute Heart Failure Patients
Brief Title: Study to Evaluate the Effectiveness of High Dose Statin Loading in Acute Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2010-0014
Record Dates: First submitted 2010-05-18; First posted 2010-05-21 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- atorvastatin 80mg (Experimental)
  Interventions: Drug: statin
- conventional therapy (for heart failure) (Active Comparator)
  Interventions: Drug: statin

INTERVENTIONS:
Drug: statin — 1. adding atorvastatin 80mg, po on day (1 to 3) acute heart failure therapy
  2. acute heart failure therapy

SUMMARY:
This is a prospective, single-center, randomized, controlled, open-label, pilot study to evaluate the effectiveness of high dose statin loading in acute heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea at rest or minimal activity
* Tachypnea (respiratory rate > 20/min) or rales or pulmonary edema on chest X-ray

Exclusion Criteria:

* Acute coronary Syndrome
* Hospitalization plan for PTCA or CABG
* Cardiogenic shock (Systolic Blood Pressure < 80mmHg)
* Uncontrolled hypertension (Systolic Blood Pressure > 180mmHg)
* Allergy, adverse drug reaction, hypersensitivity to statin
* Troponin > 5 times upper limit of normal (ULN)
* Creatinine kinase-MB level > 3 times ULN
* AST, ALT > 3 times ULN or acute hepatitis
* Current or past history of muscle disease, rhabdomyolysis
* Life expectancy < 6 months (e.g. metastatic malignancy, liver cirrhosis)
* Pregnancy or women at age of childbearing potential

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
hsCRP levels | at hospital day #4
  to investigate the effect of high dose statin loading on the change of serum NT-proBNP, hsCRP levels in patients with acute heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Min Kang, Study Director — Severance Cardiovascular hospital, Yonsei University College of Medicine; Hui-Nam Pak, Principal Investigator — Severance Cardiovascular hospital, Yonsei University College of Medicine; Boyoung Joung, Principal Investigator — Severance Cardiovascular hospital, Yonsei University College of Medicine; Sungha Park, Principal Investigator — Severance Cardiovascular hospital, Yonsei University College of Medicine
Locations (1):
- Severance Cardiovascular hospital, Yonsei University College of Medicine, Seoul, South Korea